CLINICAL TRIAL: NCT02036008
Title: Gadofosveset Trisodium (Ablavar, Gdfos) in Distinguishing Hemangiomas and Metastases: A Prospective Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 153-2013
Record Dates: First submitted 2013-10-30; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Cancer; Metastases; Liver Neoplasms
Keywords: Liver metastases; MRI; Contrast Agents
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — gadofosveset trisodium; gadobutrol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liver MRI with EcGd and with Gdfos (Other): All participants will receive two contrast-enhanced MRI studies of the liver: one with gadofosveset trisodium (Gdfos) and one with gadobutrol (EcGd) at a dose of 0.1 mL/kg body mass up to 10 mL.
  Interventions: Other: Liver MRI with Gdfos; Other: Liver MRI with EcGd

INTERVENTIONS:
Other: Liver MRI with Gdfos — Participants will receive Gdfos at a dose of 10 mL of 0.25mmol/mL. This will be administered automatically using an MRI-compatible power injector, as a bolus through an intravenous line placed in an antecubital vein at a rate of 1.5 mL/s followed by 25 mL of 0.9% saline flush.
  Participants will be imaged using a 3.0 T MRI scanner with an 8 channel body phased array coil utilized covering the entire liver. Images of the liver will be obtained including: axial precontrast phase, axial arterial phase, axial portovenous phase, axial 5 minute delayed phase, axial 10 minute delayed phase, axial 20 minute delayed phase.
  This study will be performed within 4 weeks of the MRI study with EcGd.
  Other Names: Gadofosveset trisodium (Gdfos)
Other: Liver MRI with EcGd — Participants will receive a liver MRI with EcGd as per clinical institutional protocol.
  Participants will receive EcGd at a dose of 0.1 mL/kg body mass up to 10 mL. This will be administered automatically using an MRI-compatible power injector, as a bolus through an intravenous line placed in an antecubital vein at a rate of 1.5 mL/s followed by 25 mL of 0.9% saline flush.
  Participants will be imaged using a 3.0 T MRI scanner with an 8 channel body phased array coil utilized covering the entire liver. Images of the liver will be obtained including: axial precontrast phase, axial arterial phase, axial portovenous phase, axial 5 minute delayed phase, axial 10 minute delayed phase, axial 20 minute delayed phase. Additional noncontrast images will be obtained as per institutional protocol, including diffusion weighted imaging, in/out of phase imaging, and T2 weighted imaging.
  Other Names: gadobutrol (Gadovist, EcGd)

SUMMARY:
The purpose of this study is to determine if Gadofosveset Trisodium (Gdfos, Ablavar) is a useful magnetic resonance imaging (MRI) contrast agent in accurately diagnosing liver metastases compared to the standard agent gadobutrol (EcGd, Gadovist).

DETAILED DESCRIPTION:
The proposed study will be a single centre, prospective trial comparing the sensitivity and specificity of using Gadofosveset Trisodium (Gdfos, Ablavar) as the MRI contrast agent as compared to gadobutrol (EcGd, Gadovist).

The study population will include cancer patient's referred for an MRI study of the liver to rule out metastases. Those who meet the inclusion/exclusion criteria will their routine (clinical) MRI of the liver with EcGd. They will also receive an additional MRI with Gdfos within 4 weeks of the original study.

The patient data will be anonymized and the imaging will be read by radiologists and radiology residents and comparison will be made between the diagnostic accuracy of the EcGd-enhanced study and the Gdfos-enhanced study.

ELIGIBILITY:
Inclusion Criteria:

* known cancer
* referred for MRI of liver to rule out metastases
* has focal liver lesions
* age > 18 yo

Exclusion Criteria:

* contraindication to MRI or MR contrast agents
* pregnancy
* unable to obtain all sequences and/or acceptable quality imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Reader diagnostic accuracy using Gdfos vs. EcGd compared to gold standard | Participants will receive both Gdfos and EcGd study within 4 weeks of each other. Radiologist reading for the study will be done up to 52 weeks after first MRI has been performed.
  Three blinded radiologists of different training levels will read the MRI liver studies done using Gdfos and EcGd and the results of this will be compared to a gold standard (either pathology from surgery or biopsy or long-term follow-up). The diagnostic accuracy of Gdfos vs. EcGd will be compared using area under receiver operating characteristic (ROC) curves (with correction for correlation and clustering).

SECONDARY OUTCOMES:
Inter-reader variability for EcGd-enhanced vs. Gdfos-enhanced imaging | Participants will receive both Gdfos and EcGd study within 4 weeks of each other. Radiologist reading for the study will be done up to 52 weeks after first MRI has been performed.
  Three blinded radiologists of different training levels will read the MRI liver studies done using Gdfos and EcGd and the results of this will be compared to a gold standard (either pathology from surgery or biopsy or long-term follow-up). The difference in accuracy will be compared between readers using kappa statistics.
Reader diagnostic accuracy of EcGd-enhanced imaging vs. Gdfos-enhanced imaging compared to gold standard (subgroup analysis for small lesions less than or equal to 1cm) | Participants will receive both Gdfos and EcGd study within 4 weeks of each other. Radiologist reading for the study will be done up to 52 weeks after first MRI has been performed.
  Subgroup analysis for small lesions. The same analysis will be done with only a subgroup of small lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Milot, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Milot L, Haider M, Foster L, McGregor C, Law C. Gadofosveset trisodium in the investigation of focal liver lesions in noncirrhotic liver: Early experience. J Magn Reson Imaging. 2012 Sep;36(3):738-42. doi: 10.1002/jmri.23650. Epub 2012 Apr 5. PMID 22488745